CLINICAL TRIAL: NCT03517007
Title: The DETOURS Trial: De-escalating Empiric Treatment: Opting Out of Rx for Selected Patients With Suspected Sepsis - Opt-Out Protocol Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00092813
Record Dates: First submitted 2018-05-03; First posted 2018-05-07 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2020-08

CONDITIONS: Antibiotic Stewardship
Keywords: antibiotic de-escalation; sepsis; antimicrobial stewardship
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opt-Out Protocol (Experimental): Should an eligible patient pass the safety screen and be randomized to the intervention arm of the trial, the designated pharmacist will approach the patient's primary provider in charge of antibiotic decision-making The pharmacist will inform the provider the patient's antibiotics can be de-escalated unless the provider opts out.
  Interventions: Other: Opt-Out Protocol
- Standard of Care (No Intervention): Provider continues routine, standard of care on the patient.

INTERVENTIONS:
Other: Opt-Out Protocol — Should an eligible patient pass the safety screen and be randomized to the intervention arm of the trial, the designated pharmacist will approach the patient's primary provider in charge of antibiotic decision-making The pharmacist will inform the provider the patient's antibiotics can be de-escalated unless the provider opts out.
  Arms: Opt-Out Protocol

SUMMARY:
The objective of this study is to implement an opt-out protocol to guide appropriate de-escalation of antibiotics in qualifying patients. The protocol, determined over the course a year with the help of a large, well-rounded expert panel, will be used by pharmacists to recommend de-escalation of antibiotics to hospital providers. Providers can then decide whether or not to follow the recommendation in determining the best treatment pathway for his or her patient.

ELIGIBILITY:
Inclusion Criteria:

* Blood culture preliminary results that indicate no growth as of 48-96 hours. (Exception: Patients with a single positive blood culture for coagulase negative Staphylococcus and no central line in place will also be included).
* Still on broad spectrum antibiotic therapy after 48-96 hours.

Exclusion Criteria:

* Adult patients who are located in ICU wards.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 762 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
Overall inpatient plus post-discharge antibacterial Days of Therapy (DOT) as measured by data collection | 30 days post-randomization
  Overall inpatient plus post-discharge antibacterial Days of Therapy (DOT) as measured by data collection

SECONDARY OUTCOMES:
Distributions of DOOR | up to 2 years
  DOOR is defined as Desirability of Outcome Ranking, from Alive being a rank of 1 to Death being a rank of 6. DOOR will be applied to collected patient data.
Negative outcomes as measured by individual clinical outcome components in the DOOR | 30 days post-randomization
  Negative outcomes as measured by individual clinical outcome components in the DOOR
Negative outcomes as measured by length of hospital stay | 30 days post-randomization
  Negative outcomes as measured by length of hospital stay
Negative outcomes as measured by re-initiation of antibiotic therapy after greater than 48 hours with no antibiotics | 30 days post-randomization
  Negative outcomes as measured by re-initiation of antibiotic therapy after greater than 48 hours with no antibiotics
Negative outcomes as measured by number of days patient has a central line | 30 days post-randomization
  Negative outcomes as measured by number of days patient has a central line
percent of eligible patients with antibiotic de-escalation | 5 days from initial date of suspected sepsis
  percent of eligible patients with antibiotic de-escalation
Number of patients in whom the safety screen was applied | within 3 days (96 hours) of initial date of suspected sepsis
  for patients eligible for assessment of de-escalation
Number of patients the safety screen excluded from the opt-out procedure | within 3 days (96 hours) of initial date of suspected sepsis
  for patients eligible for assessment of de-escalation
number of eligible patients in whom the opt-out procedure was applied | within 3 days (96 hours) of initial date of suspected sepsis
  for patients eligible for assessment of de-escalation
number of eligible patients in whom the prescriber chose to opt-out | within 3 days (96 hours) of initial date of suspected sepsis
  for patients eligible for assessment of de-escalation
prescriber type | within 3 days (96 hours) of initial date of suspected sepsis
  for prescribers who chose to opt out
prescribers' reported rationale for opting out | within 3 days (96 hours) of initial date of suspected sepsis
  for prescribers who chose to opt out
Percent of subjects who received an infectious disease consultation after implementation of the Opt-Out Protocol | 30 days post-randomization
  Percent of subjects who received an infectious disease consultation after implementation of the Opt-Out Protocol
Days of therapy for specific sub-groups of patients, including patients whose physicians elected to opt-out of the intervention | 30 days post-randomization
  .Days of therapy for specific sub-groups of patients, including patients whose physicians elected to opt-out of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Rebekah Moehring, MD, MPH, Principal Investigator — Duke University
Locations (10):
- United States (10):
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Piedmont Newnan Hospital, Newnan, Georgia
  - Harvard Brigham and Women's Hospital, Boston, Massachusetts
  - Duke University, Durham, North Carolina
  - Southeastern Regional Medical Center, Lumberton, North Carolina
  - Iredell Health System, Statesville, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Pennsylvania Presbyterian Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moehring RW, Yarrington ME, Warren BG, Lokhnygina Y, Atkinson E, Bankston A, Collucio J, David MZ, Davis AE, Davis J, Dionne B, Dyer AP, Jones TM, Klompas M, Kubiak DW, Marsalis J, Omorogbe J, Orajaka P, Parish A, Parker T, Pearson JC, Pearson T, Sarubbi C, Shaw C, Spivey J, Wolf R, Wrenn RH, Dodds Ashley ES, Anderson DJ; Centers for Disease Control and Prevention's Prevention Epicenters Program. Evaluation of an Opt-Out Protocol for Antibiotic De-Escalation in Patients With Suspected Sepsis: A Multicenter, Randomized, Controlled Trial. Clin Infect Dis. 2023 Feb 8;76(3):433-442. doi: 10.1093/cid/ciac787. PMID 36167851
- [Background] Yarrington ME, Moehring RW, David MZ, Hamilton KW, Klompas M, Rhee C, Hsueh K, Ashley ED, Sinkowitz-Cochran RL, Ryan M, Anderson DJ; DETOURS Expert Panel of the CDC Prevention Epicenters Program. A modified Delphi approach to develop a trial protocol for antibiotic de-escalation in patients with suspected sepsis. Antimicrob Steward Healthc Epidemiol. 2021 Nov 8;1(1):e44. doi: 10.1017/ash.2021.205. eCollection 2021. PMID 36168480